CLINICAL TRIAL: NCT02482181
Title: Diffusion Weighted Magnetic Resonance Imaging for the Characterization of Solitary Pulmonary Lesions
Acronym: DWIMRICSPL
Status: Completed | Type: Observational
Sponsor: ÇAĞLAYAN ÇAKIR (Other)
Responsible Party: Sponsor-Investigator, ÇAĞLAYAN ÇAKIR, Director,Clinical Research, Trakya University
Organization: Trakya University (Other)
Other Study IDs: TRAKYA22
Record Dates: First submitted 2015-06-19; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Thorax Cancer
Keywords: diffusion weighted magnetic resonance imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study, is to investigate the value of diffusion weighted imaging on the differential diagnosis of solitary pulmonary lesions.

DETAILED DESCRIPTION:
When a patient is diagnosed with a lung lesion, the differential diagnosis is important, since the treatment is determined by the lesion character. The goal in the evaluation of solitary pulmonary lesions is to distinguish malignant lesions from benign lesions in as non-invasive a manner as possible. As computed tomography is widely used, the diagnosis of solitary pulmonary lesions has become easier. The size, features of the edges, shape, internal structure (calcification, fat content, cavitation, etc.), density, satellite nodule, growth rate and contrast involvement of the lesion are important properties which help to distinguish benign lesions from malignant ones. However, as the distinction is not absolute at all times, other imaging methods such as positron emission tomography and magnetic resonance are preferred. The importance of this issue is the high five-year survival rate in early-diagnosed lung cancer cases.

Diffusion is the randomized microscopic motion of water molecules. It is known that diffusion is a sensitive parameter of tissue characterization at a microscopic level. Nowadays, diffusion is measured in vivo with diffusion weighted MRI and ADC measurements.

Diffusion weighted imaging has a wide use on oncologic patients for the purpose of diagnosis. In addition, it is used in the distinction of acute cerebral infarction and epidermoid or arachnoid cysts. Recently, it has also been used in the characterization of cystic or solid lesions in the thoracic cavity. In this study, the investigators aimed to evaluate the accuracy of differentiation of solitary pulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients had a solitary pulmonary nodule or mass.

Exclusion Criteria:

-

Ages: 20 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Magnetic resonance imaging (MRI) was applied to a total of 46 patients between January 2011 and July 2011, who presented.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
On diffusion weighted images, the signal intensities of the lesions were visually compared to the SI of the thoracic spinal cord using a 5-point scale. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: HAKAN GENÇHELLAÇ, MD, Study Director — TURKEY,EDİRNE ,TRAKYA UNİVERSİTY HOSPİTAL
Locations (1):
- Trakya University Hospital, Edi̇rne, Turkey (Türkiye)

REFERENCES:
- [Derived] Cakir C, Genchellac H, Temizoz O, Polat A, Sengul E, Duygulu G. Diffusion Weighted Magnetic Resonance Imaging for the Characterization of Solitary Pulmonary Lesions. Balkan Med J. 2015 Oct;32(4):403-9. doi: 10.5152/balkanmedj.2015.15663. Epub 2015 Oct 1. PMID 26740901